CLINICAL TRIAL: NCT02081222
Title: The Predictability of Intraoperative Rotational Thromboelastometry on Postoperative Bleeding and Transfusion Requirements
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, WonHo Kim, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-12-096
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Surgery for Congenital Heart Disease; Pediatric Patients
Keywords: congenital heart disease; rotational thromboelastometry; blood loss; transfusion requirements
MeSH Terms: conditions — Heart Defects, Congenital; Hemorrhage | interventions — Surgical Procedures, Operative; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients who underwent surgery for congenital heart disease: patients who underwent surgery for congenital heart disease in 2013 at Samsung Medical Center
  Interventions: Procedure: surgery for congenital heart disease with cardiopulmonary bypass

INTERVENTIONS:
Procedure: surgery for congenital heart disease with cardiopulmonary bypass — surgery for congenital heart disease with cardiopulmonary bypass

SUMMARY:
Viscoelastic hemostatic assay has been reported to be superior to predict perioperative bleeding in cardiac surgical patients compared with conventional blood coagulation test. However, the role of rotational thromboelastometry (ROTEM) in predicting perioperative bleeding and transfusion requirements in pediatric patients who undergoing surgery for congenital heart disease. Therefore, the investigators attempt to evaluate the predictability of intraoperative rotational thromboelastometry for perioperative bleeding and transfusion requirements in pediatric cardiac surgical patients by comparing with conventional coagulation test. The investigators also attempt to evaluate the correlation between ROTEM parameters, platelet count, and results of conventional coagulation test results.

DETAILED DESCRIPTION:
Viscoelastic hemostatic assay has been reported to be superior to predict perioperative bleeding in cardiac surgical patients compared with conventional blood coagulation test. However, the role of rotational thromboelastometry (ROTEM) in predicting perioperative bleeding and transfusion requirements in pediatric patients who undergoing surgery for congenital heart disease. Therefore, the investigators attempt to evaluate the predictability of intraoperative rotational thromboelastometry for perioperative bleeding and transfusion requirements in pediatric cardiac surgical patients by comparing with conventional coagulation test. The investigators also attempt to evaluate the correlation between ROTEM parameters, platelet count, and results of conventional coagulation test results.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients (< 10 years) who underwent surgery for congenital heart disease with cardiopulmonary bypass in 2013 at Samsung Medical Center

Exclusion Criteria:

* incomplete data about blood loss count or transfusion requirements during seven days after surgery

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients who underwent surgery for congential heart disease with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
postoperative blood loss | during seven days after surgery
  daily blood loss measured by chest tube drainage during seven days after surgery

SECONDARY OUTCOMES:
postoperative transfusion requirements | during seven days after surgery
  postoperative transfusion requirements during seven days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea